CLINICAL TRIAL: NCT04036994
Title: Photobiomodulation Therapy for the Management of Chemotherapy-induced Alopecia: a Randomized, Placebo-controlled Feasibility Trial
Brief Title: PBMT for the Management of CIA ( HAIRLASER )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Prof. dr. Jeroen Mebis, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19.58/ONCO19.08
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Chemotherapy-induced Alopecia; Alopecia
Keywords: photomodulation therapy; supportive cancer care; epirubicin cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms; Alopecia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment group (Active Comparator)
  Interventions: Device: Photobiomodulation therapy
- Control group (no intervention) (No Intervention)

INTERVENTIONS:
Device: Photobiomodulation therapy — All patients will undergo photobiomodulation therapy sessions three times a week for the total duration of 12 weeks starting at their last CT administration.
  Other Names: Low level laser therapy
  Arms: Experimental: Treatment group

SUMMARY:
Chemotherapy (CT) remains an important treatment modality for breast cancer patients. Unfortunately, this systemic treatment comes with many quality of life impairing complications. Chemotherapy-induced alopecia (CIA) occurs in about 65% of the patients. Hair loss due to CT is reversible, but hair regrowth requires several months to a year after CT. Currently, the only available preventive measure is based on scalp cooling. Nevertheless, this treatment has a highly variable success rate and it brings along several side effects. Photobiomodulation therapy (PBMT) is a new, preventive and therapeutic technique in the supportive care of cancer patients. It uses visible and (near)- infrared light produced by laser diodes or light-emitting diodes (LED) at a low power to stimulate tissue repair and reduce inflammation and pain. The investigator's research team demonstrated already that PBMT can prevent oral mucositis and acute radiodermatitis. The aim of this project is to explore the use of PBMT in the management of CIA. Results of this project will lead to an improvement of the patients' quality of life after CT.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature.
* Age 18 years or above
* Female
* Use of a wig for at least 2 hours a day
* Able to read and converse in Dutch
* Skin type I to IV on the Fitzpatrick Skin Type Scale
* Diagnosis of non-invasive (stage 0) or invasive (stage 1, 2 and 3A) breast adenocarcinoma.
* Treatment with neoadjuvant (preoperative) or adjuvant (postoperative) chemotherapy: anthracycline and taxane containing (paclitaxel or docetaxel) chemotherapy regimen.
* Diagnosed with CIA grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE)
* Have no documented or observable psychiatric or neurological disorders that might interfere with study participation (e.g., dementia or psychosis).

Exclusion Criteria:

* Metastatic disease
* Severe or unstable cardio- respiratory or musculoskeletal disease
* Pregnancy
* Presence of cognitive impairment that might impact study outcomes
* Previously (before start of chemotherapy) diagnosed with a hair loss condition
* Receiving scalp cooling during chemotherapy
* Active infection on the scalp
* Chronic dermatologic condition (e.g. eczema, psoriasis, infection)
* Take any of the following medications for 6 months prior to initiation of the study: minoxidil, finasteride (or any other 5α-reductase inhibitor medications), medications with anti-androgenic properties (e.g. cyproterone, spironolactone, ketoconazole, flutamide and bicalutamide)n medications that can potentially cause hypertrichosis (ciclosporin, diazoxide, phenytoin and psoralens), and oral glucocorticoids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | Baseline
  A mechanical visual analogue scale (VAS) will be used to evaluate the patients' hair regrowth based on photographs taken at the four time points. The patients will be asked to indicate their subjective experience of hair regrowth. This score is associated with a certain score, in which 0 = 'total baldness' and 10 = 'full scalp coverage'.
visual analogue scale (VAS) | Month 1
  A mechanical visual analogue scale (VAS) will be used to evaluate the patients' hair regrowth based on photographs taken at the four time points. The patients will be asked to indicate their subjective experience of hair regrowth. This score is associated with a certain score, in which 0 = 'total baldness' and 10 = 'full scalp coverage'.
visual analogue scale (VAS) | Month 2
  A mechanical visual analogue scale (VAS) will be used to evaluate the patients' hair regrowth based on photographs taken at the four time points. The patients will be asked to indicate their subjective experience of hair regrowth. This score is associated with a certain score, in which 0 = 'total baldness' and 10 = 'full scalp coverage'.
visual analogue scale (VAS) | Month 3
  A mechanical visual analogue scale (VAS) will be used to evaluate the patients' hair regrowth based on photographs taken at the four time points. The patients will be asked to indicate their subjective experience of hair regrowth. This score is associated with a certain score, in which 0 = 'total baldness' and 10 = 'full scalp coverage'.

SECONDARY OUTCOMES:
EORTC QLQ-C30 Quality of life questionnaire | Baseline
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
EORTC QLQ-C30 Quality of life questionnaire | Month 1
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
EORTC QLQ-C30 Quality of life questionnaire | Month 2
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
EORTC QLQ-C30 Quality of life questionnaire | Month 3
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
QLQ-BR23 Quality of life questionnaire | Baseline
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
QLQ-BR23 Quality of life questionnaire | Month 1
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
QLQ-BR23 Quality of life questionnaire | Month 2
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
QLQ-BR23 Quality of life questionnaire | Month 3
  A validated questionnaire of the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module
Patient global satisfaction numerical rating scale | Month 3
  The patients' global satisfaction with the PBMT/sham therapy will be evaluated using a numerical rating scale (NRS) from 0 (minimum score) to 10 (maximum score)

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, prof. dr., Principal Investigator — Jessa Hospital; Joy Lodewijckx, drs., Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lodewijckx J, Robijns J, Claes M, Pierson M, Lenaerts M, Mebis J. The use of photobiomodulation therapy for the management of chemotherapy-induced alopecia: a randomized, controlled trial (HAIRLASER trial). Support Care Cancer. 2023 Apr 15;31(5):269. doi: 10.1007/s00520-023-07743-1. PMID 37060420